CLINICAL TRIAL: NCT05161702
Title: Increased Inflammation-resolving Activity by Omega-3 Monoglycerides in Peripheral Blood Mononuclear Cells (PBMC).
Acronym: PBMC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SCF Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: PBMC
Record Dates: First submitted 2021-12-15; First posted 2021-12-17 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Resolution of Inflammation; Reduction of Cell Proliferation
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MAG-SPM treatment on isolated PBMC cells — Cells are isolated form the participant's blood donation (4x 10mL k2EDTA tubes per participant) and maintained in culture with LPS, a pro-inflammatory and pro-proliferative agent. Then, PBMC are separated in two, one half treated with MAG-SPM and the other half remains with LPS only. Proliferative activities are measured and compared in both cell dish.
Other: Isolated PBMC cells without treatment. — Cells are isolated form the participant's blood donation (4x 10mL k2EDTA tubes per participant) and maintained in culture with LPS, a pro-inflammatory and pro-proliferative agent. Then, PBMC are separated in two, one half treated with MAG-SPM and the other half remains with LPS only. Proliferative activities are measured and compared in both cell dish.

SUMMARY:
The purpose of this biological study is to provide Dr. Samuel Fortin's laboratory with a continuous supply of blood mononuclear cells (PBMCs) so that he can pursue research on the potential beneficial effects of monoglyceride omega-3 fatty acids on the resolution of inflammation.

DETAILED DESCRIPTION:
The biological activity of omega-3 fatty acids requires selective oxidation by lipoxygenase (LOX) enzymes in the human body to form SPM (Specialized Pro-resolving Mediators). The formulations based on omega-3 monoglyceride (MAG-Omega-3) currently marketed by SCF Pharma have been optimized so as not to interfere with this natural metabolism process in the human body. It has already been shown that the antiproliferative activity of docosapentaenoic acid (or omega-3 ADP) can be increased tenfold when it is pre-metabolized using a LOX enzyme from soybean (C. Morin et al. PLEFA (2013) 203-213). This antiproliferative potential may play a key role in the mechanisms of inflammation resolution.

We now want to develop a new line of high performance products by pre-metabolizing MAG-Omega-3 in the form of SPM monoglycerides (MAG-SPM) using the LOX enzyme from soy. The potential for resolving inflammation by MAG-SPM can be measured by cell proliferation assays. To perform these tests, cells of the PBMC type must be isolated from the blood of donors and maintained in culture in the presence of an inflammatory agent (LPS) which induces their proliferation (C. Morin et al. European Journal of Pharmacology 807 (2017)) 205-211). Next, the reduction in proliferation induced by MAG-SPM is quantified and then compared with that of cells not treated with MAG-SPM. This type of test requires a large amount of fresh cells, and therefore, a source of blood sample supply.

This research project is divided into two parts: 1) A protocol for collecting blood samples; 2) A cell proliferation test protocol to demonstrate the activity of MAG-SPM in the resolution of inflammation. This protocol covers the first part of this research project.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged of at least 18 years old.

Exclusion Criteria:

* Participant who use omega-3 supplements and / or anti-inflammatory medication such as, but not limited to - Aspirin, Ibuprofen (Motrin, Advil), Celecoxib (Celebrex), diclofenac (Cambia, Cataflam, Voltaren ) within 7 days of day 1 of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult blood donors
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of PBMC cells count | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel P Fortin, PhD, Principal Investigator — SCF Pharma
Locations (1):
- SCF Pharma, Rimouski, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No